CLINICAL TRIAL: NCT02498743
Title: Effect of Television Cartoons in Patients Younger Than 3.5 Years During Echocardiography.A Prospective Randomized Study
Brief Title: Effect of Television Cartoons in Patients Younger Than 3.5 Years During Echocardiography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana (Other)
Responsible Party: Principal Investigator, Francisco Sánchez Ferrer, MD, Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2015-01
Record Dates: First submitted 2015-07-10; First posted 2015-07-15 (Estimated); Last update posted 2015-07-15 (Estimated); Status verified 2015-07

CONDITIONS: Echocardiography; Pediatrics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention group with television (Experimental): Animated cartoons with sound were reproduced during the echocardiography
  Interventions: Procedure: echocardiography; Behavioral: Watching Animated cartoons
- control group with usual care (No Intervention): Echocardiography was performed by using the distractions available at the time of test.

INTERVENTIONS:
Procedure: echocardiography — TV was connected to display the cartoon video during the echocardiography: the episode number 125 of 'Dora the Explorer': 'Baby Winky Goes Home!' was reproduced during the echocardiography.
  Arms: Intervention group with television
Behavioral: Watching Animated cartoons
  Arms: Intervention group with television

SUMMARY:
The objective of this study is analyze the influence of TV entertainment in children less than 3 years of age during echocardiography in order to achieve a complete and accurate test.

This is an experimental study in children with suspected congenital or acquired cardiac disease. An examination room was prepared with a TV on the ceiling that was positioned in a way that would provide unobstructed viewing for children during the echocardiography procedure.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients who were referred to pediatric cardiology consultation.
* Patients younger than 3.5 years.
* Signed informed consent by parents.

Exclusion Criteria:

* No signed informed consent by parents.

Ages: 6 Months to 43 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 58 (Actual)
Dates: Start 2015-02; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Echocardiography time | procedure
  Time used to perform the Echocardiography
Quality of technique | procedure
  The quality of echocardiography (1 poor, 2 medium, 3 high)

SECONDARY OUTCOMES:
Parents opinion | procedure
  Parents completed a questionnaire about the use of TV during the test
Parents stress | procedure
  The parent's opinion about the sensation of stress by using a scale from 0 (no stress) to 10 (so much stress
Blood pressure | procedure
  blood pressure of child

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Sanchez Ferrer, MD, Principal Investigator — Hospital San Juan de Alicante
Locations (1):
- Francisco Sánchez Ferrer, Sant Joan d'Alacant, Alicante, Spain

REFERENCES:
- [Background] Mertens L, Friedberg MK. The gold standard for noninvasive imaging in congenital heart disease: echocardiography. Curr Opin Cardiol. 2009 Mar;24(2):119-24. doi: 10.1097/HCO.0b013e328323d86f. PMID 19225295
- [Background] Mertens L, Seri I, Marek J, Arlettaz R, Barker P, McNamara P, Moon-Grady AJ, Coon PD, Noori S, Simpson J, Lai WW; Writing Group of the American Society of Echocardiography; European Association of Echocardiography; Association for European Pediatric Cardiologists. Targeted Neonatal Echocardiography in the Neonatal Intensive Care Unit: practice guidelines and recommendations for training. Writing Group of the American Society of Echocardiography (ASE) in collaboration with the European Association of Echocardiography (EAE) and the Association for European Pediatric Cardiologists (AEPC). J Am Soc Echocardiogr. 2011 Oct;24(10):1057-78. doi: 10.1016/j.echo.2011.07.014. No abstract available. PMID 21933743
- [Background] Heistein LC, Ramaciotti C, Scott WA, Coursey M, Sheeran PW, Lemler MS. Chloral hydrate sedation for pediatric echocardiography: physiologic responses, adverse events, and risk factors. Pediatrics. 2006 Mar;117(3):e434-41. doi: 10.1542/peds.2005-1445. Epub 2006 Feb 15. PMID 16481449
- [Background] American Academy of Pediatrics; American Academy of Pediatric Dentistry; Cote CJ, Wilson S; Work Group on Sedation. Guidelines for monitoring and management of pediatric patients during and after sedation for diagnostic and therapeutic procedures: an update. Paediatr Anaesth. 2008 Jan;18(1):9-10. doi: 10.1111/j.1460-9592.2007.02404.x. No abstract available. PMID 18095958